CLINICAL TRIAL: NCT06125405
Title: Study of the Telitacicept in Pediatric Patients With Frequently Relapsing or Steroid Dependent Nephrotic Syndrome
Acronym: STERN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Mao Jianhua, Professor, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STERN
Record Dates: First submitted 2023-10-24; First posted 2023-11-09 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Nephrotic Syndrome in Children; Telitacicept
Keywords: Telitacicept; Frequently Relapsing Nephrotic Syndrome; Steroid Dependent Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — telitacicept

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telitacicept group (Experimental): Weekly administration (administration time can be within 1 week + 3 days). Body weight and dosage: for subjects with body weight greater than 10kg and less than or equal to 20kg, the dose of Telitacicept is 40mg; for subjects with body weight greater than 20kg and less than or equal to 40kg, the dose of Telitacicept is 80mg; for subjects with body weight greater than 40kg and less than or equal to 60kg, the dose of Telitacicept is 120mg; for subjects with body weight greater than or equal to 60kg, the dose of Telitacicept is 160mg. Treatment duration: 52 weeks.
  Interventions: Drug: Telitacicept

INTERVENTIONS:
Drug: Telitacicept — The study duration was 52 weeks, with the experimental group receiving subcutaneous injections of Telitacicept once weekly for a total of 52 weeks.

SUMMARY:
The main objective is to evaluate the effectiveness of telitacicept in pediatric patients with frequently relapsing or steroid dependent nephrotic syndrome within the 52-week follow-up.

DETAILED DESCRIPTION:
Nephrotic syndrome(NS) is the most common glomerular disease in children. Approximately 45-50% of patients with nephrotic syndrome exhibit frequent relapses or are dependent on steroid therapy. Frequent relapses or steroid dependence in nephrotic syndrome have been challenging issues for clinicians. Long-term, repeated, and high-dose oral steroid use can lead to side effects such as obesity, delayed development, hypertension, diabetes, glaucoma, osteoporosis, and increased susceptibility to infections. The addition of traditional immunosuppressants such as cyclophosphamide and tacrolimus can cause severe and irreversible side effects. Therefore, exploring new drugs and their application protocols is particularly important. Telitacicept has a unique dual-target mechanism that can inhibit B cell maturation and differentiation at multiple stages, thereby inhibiting B cell activity. Clinical studies have confirmed its significant efficacy in various kidney diseases, such as lupus nephritis, IgA nephropathy, and adult recurrent minimal change nephrotic syndrome; moreover, it has good safety profiles.

Therefore, through this prospective, single-center, open-label clinical trial, we aim to evaluate whether telitacicept provides superior efficacy compared to existing conventional treatment regimens for childhood frequent relapse (FR) or steroid-dependent (SD) nephrotic syndrome (NS), and assess its safety profile. Our goal is to provide an optimized treatment plan for childhood FRNS or SDNS.

ELIGIBILITY:
Inclusion Criteria:

* Sensitive but frequent relapses or steroids dependence nephrotic syndrome
* Age: 2 to 18 years old
* Normal renal function: estimated glomerular filtration rate ≥90ml/ min/1.73m2
* Morning urine protein <1+ or urine protein-creatinine ratio <0.2g/g (<20 mg/ mmol) for 3 consecutive days and above when in enroll
* No rituximab was used within 6 months, no tacrolimus, mycophenolate mofetil, cyclosporine A, or cyclophosphamide was used within 3 months, no ACTH was used within 3 months prior to the enrollment

Exclusion Criteria:

* Family history of nephrotic syndrome, chronic glomerulonephritis or uremia
* Leukopenia (White Blood Cells ≤ 3.0 * 10^9 / L)
* Moderate to severe anemia (hemoglobin <9.0 g/dL)
* Thrombocytopenia (platelet count <100*10^12/L)
* Positive Hepatitis B virus serological indicators (Hepatitis B surface antigen or / and Hepatitis B virus e antigen or / and Hepatitis B core antibody), Hepatitis C virus-positive or patients with abnormal liver function (2 or more times of alamine aminotransferase or total bilirubin was exceeded the normal value, and continued to rise for 2 weeks)
* There are chronic active infections such as Epstein-Barrvirus, cytomegalovirus or Mycobacterium tuberculosis, and the usage of steroids and immunosuppressive agents may aggravate the state of an illness
* Secondary nephrotic syndrome (such as purpuric nephritis, lupus nephritis, etc.)
* Those who with hematological or endocrine system diseases as well as serious organs illness such as heart, liver or kidney
* Those who with other autoimmune diseases or primary immunodeficiencies or tumors
* Those who have participated in other clinical trials within three months prior to the enrollment
* Those who was not suitable for participating this study judged by investigator

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-10-24 (Estimated); Study Completion 2027-10-24 (Estimated)

PRIMARY OUTCOMES:
1-year relapse-free survival rate | 1-year period after enrollment
  The rate of no relapse within 1 year

SECONDARY OUTCOMES:
Relapse of nephrotic syndrome during 12 months after enrollment | 1-year period after enrollment
  Proportion of patients with one or more relapse(s) of nephrotic syndrome
Number of relapses during 12 months follow up | 1-year period after enrollment
  Number of nephrotic syndrome relapses per patient year during the 12 months period after enrollment
The first time to relapse | 1-year period after enrollment
  The first time to relapse after patients taking part in this study
Cumulative prednisone dosage (milligrams per kilogram per year) | 1-year period after enrollment
  The total dosage of prednisones from the beginning to the end of the trial
Change in hemoglobin of the patients | 1-year period after enrollment
  The changes of hemoglobin (g/L) in each follow-up during the study
Change in blood albumin of the patients | 1-year period after enrollment
  The changes of blood albumin (g/L）in each follow-up during the study
Change in renal function of the patients | 1-year period after enrollment
  The change for renal function was judged by the changes of estimated glomerular filtration rate (eGFR in ml/min/1.73m^2) in each follow-up during the study
Change in mass index (BMI) during 12-month period after enrollment | 1-year period after enrollment
  Changes in standard deviation scores for weight (Wt in kilograms), height (Ht in meters) will be combined to report body mass index (BMI in kg/m^2) during 12-month period after enrollment

OTHER OUTCOMES:
Adverse event | 1-year period after enrollment
  The number of harmful reactions and the types of adverse events during the study

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Mao, MD, Principal Investigator — Children's Hospital, Zhejiang University School of Medicine
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veltkamp F, Rensma LR, Bouts AHM; LEARNS consortium. Incidence and Relapse of Idiopathic Nephrotic Syndrome: Meta-analysis. Pediatrics. 2021 Jul;148(1):e2020029249. doi: 10.1542/peds.2020-029249. Epub 2021 Jun 30. PMID 34193618
- [Background] Eddy AA, Symons JM. Nephrotic syndrome in childhood. Lancet. 2003 Aug 23;362(9384):629-39. doi: 10.1016/S0140-6736(03)14184-0. PMID 12944064
- [Background] Filler G, Young E, Geier P, Carpenter B, Drukker A, Feber J. Is there really an increase in non-minimal change nephrotic syndrome in children? Am J Kidney Dis. 2003 Dec;42(6):1107-13. doi: 10.1053/j.ajkd.2003.08.010. PMID 14655180
- [Background] Tarshish P, Tobin JN, Bernstein J, Edelmann CM Jr. Prognostic significance of the early course of minimal change nephrotic syndrome: report of the International Study of Kidney Disease in Children. J Am Soc Nephrol. 1997 May;8(5):769-76. doi: 10.1681/ASN.V85769. PMID 9176846
- [Background] Dhillon S. Telitacicept: First Approval. Drugs. 2021 Sep;81(14):1671-1675. doi: 10.1007/s40265-021-01591-1. PMID 34463932
- [Background] Shi F, Xue R, Zhou X, Shen P, Wang S, Yang Y. Telitacicept as a BLyS/APRIL dual inhibitor for autoimmune disease. Immunopharmacol Immunotoxicol. 2021 Dec;43(6):666-673. doi: 10.1080/08923973.2021.1973493. Epub 2021 Sep 14. PMID 34519594
- [Background] Cai J, Gao D, Liu D, Liu Z. Telitacicept for autoimmune nephropathy. Front Immunol. 2023 Jun 5;14:1169084. doi: 10.3389/fimmu.2023.1169084. eCollection 2023. PMID 37342346
- [Background] Chen R, Fu R, Lin Z, Huang C, Huang W. The efficacy and safety of telitacicept for the treatment of systemic lupus erythematosus: a real life observational study. Lupus. 2023 Jan;32(1):94-100. doi: 10.1177/09612033221141253. Epub 2022 Nov 23. PMID 36416639
- [Background] Lv J, Liu L, Hao C, Li G, Fu P, Xing G, Zheng H, Chen N, Wang C, Luo P, Xie D, Zuo L, Li R, Mao Y, Dong S, Zhang P, Zheng H, Wang Y, Qin W, Wang W, Li L, Jiao W, Fang J, Zhang H. Randomized Phase 2 Trial of Telitacicept in Patients With IgA Nephropathy With Persistent Proteinuria. Kidney Int Rep. 2022 Dec 29;8(3):499-506. doi: 10.1016/j.ekir.2022.12.014. eCollection 2023 Mar. PMID 36938094
- [Background] Li S, Ding L, Yang YJ, Yang XD. Telitacicept for minimal change disease. Kaohsiung J Med Sci. 2023 Jul;39(7):748-749. doi: 10.1002/kjm2.12719. No abstract available. PMID 37440467